CLINICAL TRIAL: NCT06035536
Title: A Multi-Center, Randomized Controlled Clinical Investigation Evaluating Wound Closure With Symphony™ Versus Standard of Care in the Treatment of Non-Healing Diabetic Foot Ulcers
Brief Title: Clinical Study Evaluating Symphony™ Versus Standard of Care in the Treatment of Non-Healing Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aroa Biosurgery Limited (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AROA 003
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Foot Ulcer; Chronic Foot Ulcer
Keywords: Extracellular matrix; Regenerative medicine; Leg ulcer; Diabetes Mellitus; Diabetic Angiopathies; Diabetes Complications
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Leg Ulcer; Diabetes Mellitus; Diabetic Angiopathies; Diabetes Complications

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Symphony™ treatment (Experimental): Arm receives an application of Symphony™ treatment and appropriate Off-loading.
  Interventions: Device: Symphony™ plus Off-loading
- Standard of Care (SOC) treatment (Active Comparator): Arm receives an application of SOC comprising of calcium alginate Fibracol dressing and appropriate Off-loading.
  Interventions: Device: Wound Dressing comprising of calcium alginate Fibracol

INTERVENTIONS:
Device: Symphony™ plus Off-loading — Application of Symphony™
  Arms: Symphony™ treatment
Device: Wound Dressing comprising of calcium alginate Fibracol — Application of Wound Dressing comprising of calcium alginate Fibracol.
  Arms: Standard of Care (SOC) treatment

SUMMARY:
The study will evaluate the safety and performance of Symphony™ versus Standard of Care (SOC) in the treatment of chronic non-healing diabetic foot ulcers (DFU) after 12 weeks of treatment.

DETAILED DESCRIPTION:
About 120 subjects will take part in this study. Subjects with a Wagner Grade 1 or 2 Diabetic Foot Ulcers will be randomized at a ratio of 1:1 to one of the two treatment groups at the time of completion of screening to either Symphony™ treatment or Standard of Care (SOC) treatment groups.

Following initial enrolment, eligible subjects will then undergo:

* A screening phase consisting of 14 days to determine eligibility.
* Eligible subjects will then undergo a treatment phase involving weekly treatment and evaluations for up to 12 weeks.
* Subjects that heal will undergo a follow-up phase that includes 1 visit (Healing Confirmation Visit), 2 weeks from initial healing.
* If the subject does not heal, they will exit at Week 13, End of Study visit.

Both treatment groups will receive accepted routine procedures being part of SOC, including offloading of the DFU (removable cast boot or total contact casting [TCC] if the subject's foot is too large for a removable cast boot), appropriate sharp or surgical debridement, and infection management.

In addition to what is noted above, Group 1 will receive a weekly application of Symphony™ and Group 2 will receive SOC comprising of calcium alginate Fibracol dressing. Both Groups will have a silicone non-adherent dressing (MepitelTM or equivalent), a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll, compressive wrap and Coban (Threeflex 3layer or equivalent) applied.

ELIGIBILITY:
Inclusion Criteria:

* 1. At least 18 years old, inclusive.
* 2. Presence of a DFU, Wagner Grade 1 or 2 (see Appendix B for definitions), extending through the dermis provided it is below the medial aspect of the malleolus.
* 3. The index ulcer (ulcer to be evaluated in the study) will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
* 4. Index ulcer has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
* 5. Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
* 6. Within 3 months of SV1, adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
* 7. The target ulcer has been offloaded for at least 14 days, prior to TV1.
* 8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* 9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
* 10. Subjects must have read and signed the IRB approved ICF before screening procedures are performed.

Exclusion Criteria:

* 1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes
* 2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer
* 3. Index ulcer is overtly infected (i.e., purulent drainage)
* 4. Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study
* 5. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1
* 6. History of radiation at the ulcer site (regardless of time since last radiation treatment)
* 7. Index ulcer has been previously treated or will need to be treated with any prohibited therapies
* 8. Subjects with a previous diagnosis of HIV or Hepatitis C
* 9. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment
* 10. Osteomyelitis or bone infection of the affected foot as verified by xray within 30 days prior to the first screening visit. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision)
* 11. Subject is pregnant or breast-feeding
* 12. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within last 90 days
* 13. Subjects with end stage renal disease as evidenced by a serum creatinine ≥3.0 mg/dL within 6 months of enrollment
* 14. Presence of acute Charcot Neuroarthropathy to the affected limb
* 15. Index ulcer that has reduced in area by 30% or more after 14 days of SOC from SV1 to the TV1/Randomization visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Percentage of index ulcers healed at 12 weeks | 12 weeks
  Percentage of index ulcer defined as 100% re-epithelialization within 12 weeks

SECONDARY OUTCOMES:
Time to heal within 12 weeks | 12 weeks
  Time to heal of index ulcer defined as 100% re-epithelialization within 12 weeks
Percentage area reduction at 12 weeks | 12 weeks
  Area reduction percentage of ulcer at 12 weeks
Changes in wound quality of life (per W-QoL) | after 12 weeks
  Changes in wound quality of life (W-QoL) using the W-QoL short questionnaire administered on Study Visit 1 (as a baseline) and after 12 weeks of treatment (End of Study Visit) normalized to a single value. Each item is scored on a 5-point Likert scale from 0 (not at all) to 4 (very much).
Change in pain levels during the clinical investigation | 12 weeks
  Change in subject-reported pain levels using the 0-10 Numeric Pain Rating Scale at each weekly visit. On the numerical pain scale, the number 0 represents "no pain" and the number 10 represents "the worst possible pain".

OTHER OUTCOMES:
Product wastage (Symphony only) | 12 weeks
  Product wastage (applies only to DFUs treated with Symphony). Area of Symphony device; wound area at time of application based on digital planimetry imaging of area. Percentage wastage: (Area of DFU - area of Symphony/area of DFU) x 100.
Cost to closure (both treatment groups; all wounds, and only closed wounds) | 12 weeks
  Costs for all wounds per treatment group, and cost of healed wounds only per treatment group. Final values are cost per wound.

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD PhD, Study Chair — Keck School of Medicine
Locations (11):
- United States (11):
  - LA Foot and Ankle, Los Angeles, California
  - Clemente Clinical Research Inc., Los Angeles, California
  - Bay Area Foot Care, San Francisco, California
  - Doctor's Research Network, Miami, Florida
  - Barry University Clinical Research, Tamarac, Florida
  - Curalta Foot and Ankle, Westwood, New Jersey
  - Foot and Ankle Specialists of the Mid-Atlantic, Gastonia, North Carolina
  - Lower Extremity Institute for Research and Therapy, Boardman, Ohio
  - Martin Foot and Ankle, York, Pennsylvania
  - Perfizien Clinical Research, Houston, Texas
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No